CLINICAL TRIAL: NCT03287778
Title: Randomized Controlled Trial of Pyridoxine for Tardive Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1500
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Tardive Dyskinesia; Antipsychotic Agents
Keywords: Pyridoxine; Vitamin B6; Neurologic Manifestations; Involuntary Movements; Movement Disorder; Dyskinesias; Physiological Effects of Drugs; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Signs and Symptoms
MeSH Terms: conditions — Tardive Dyskinesia; Neurologic Manifestations; Dyskinesias; Movement Disorders; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Signs and Symptoms | interventions — Pyridoxine; Vitamin B 6; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyridoxine (Active Comparator): Pyridoxine will be administered in dosages of 200 mg with a maximum dose of 400 mg.
  Interventions: Dietary Supplement: Pyridoxine
- Placebo (Placebo Comparator): Matching placebos will be administered for each active drug.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pyridoxine — Max dose of 400 mg QD PO
  Other Names: Vitamin B6
  Arms: Pyridoxine
Dietary Supplement: Placebo — Matching placebos will be administered.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Purpose: Tardive dyskinesia (TD) is a involuntary movement disorder that can occur following long term treatment with antipsychotic medications and for which few treatment options exist. This study will test the efficacy of pyridoxine (also known as vitamin B6) for TD. This will be an 8 week double-blind, placebo-controlled, randomized trial measuring the effect of pyridoxine 400 mg/day on the severity of involuntary muscle movements in people who meet Schooler-Kane criteria for TD.

Participants: Approximately 50 subjects will be recruited from the UNC Schizophrenia Treatment and Evaluation Program (STEP) and other local psychiatric clinics.

Procedures (methods): Symptoms of TD will be assessed using the Abnormal Involuntary Movement Scale (AIMS). Pharmacological Intervention: All participants who meet entry criteria will be randomized to one of two treatment groups: pyridoxine or placebo.

DETAILED DESCRIPTION:
Overview of Procedures: All procedures will be conducted at either the University of North Carolina Hospitals in Chapel Hill, or at the North Carolina Psychiatric Research Center (NCPRC), a specialized program of the University of North Carolina Center for Excellence in Community Mental Health, in Raleigh.

Screening: During the initial clinic visit and after providing written informed consent, prospective subjects' psychiatric and medical histories will be reviewed, physical exams conducted, demographics and vital signs obtained, and blood and urine collected. The Structured Clinical Interview for DSM-V, the Columbia Suicide Severity Rating Scale (C-SSRS), and the Clinical Global Impressions-Severity (CGI-S) will be used to evaluate psychopathology. Involuntary muscle movements will be assessed using the Abnormal Involuntary Movement Scale (AIMS). The AIMS exam will be video recorded. Other neurological side effects of antipsychotic medications will be assessed using the Barnes Akathisia Scale (BARS) and Simpson-Angus Scale (SAS).

The baseline visit will be scheduled within 28 days of the screening visit. Vital signs and weight will be measured. A blood test to measure baseline pyridoxine level will be collected. A battery of assessments will be administered including the Clinical Global Impressions-Severity (CGI-S), the Alcohol Use Scale, Substance Use Scale, Brief Psychiatric Rating Scale (BPRS), Columbia Suicide Severity Rating Scale (C-SSRS), AIMS (video recorded), BARS, and SAS.

At the completion of the baseline visit, subjects who continue to meet study inclusion criteria will be randomized to one of two treatment groups (pyridoxine or placebo). Subjects assigned to the pyridoxine group will receive 200 mg per day for one week and then 400 mg per day, as tolerated, for the remainder of the study. Subjects assigned to the placebo group will receive matching placebo capsules.

After study enrollment, subjects will be scheduled for Week 1 and Week 2 study visits. The purpose of these visits will be to assess medication management (i.e., adverse events/side effects, adherence), collect vital signs, assess current psychiatric status, and assess neurological symptoms using the AIMS (video recorded), BARS, and SAS. The CGI-S will be performed at both Week 1 and Week 2, however, the C-SSRS will be completed at Week 2 only.

Study visit at Week 4 and end-of-study visit at Week 8 will be similar to Week 2, with the addition of the BPRS, Substance Use Scale and Alcohol Use Questionnaire. A blood test to measure pyridoxine levels will also be collected during these visits. Study drug is discontinued at the Week 8 visit.

A follow-up visit at Week 10, two weeks after stopping the treatment, will consist of assessing for adverse events/side effects, collecting vital signs, administrating the CGI-S and C-SSRS, and performing the AIMS (video recorded), BARS, and SAS. The follow-up visit will help determine whether the potential benefits of pyridoxine for TD may continue after treatment is discontinued.

Vital signs, adverse events, and side effects will be obtained at all in-person study visits. Blood collection and laboratory testing will be done at Screening, Baseline, Week 4, and Week 8 .

ELIGIBILITY:
Inclusion Criteria:

* Meet Schooler - Kane criteria for TD (at least one muscle group is rated at "moderate" severity or at least two muscle groups are rated at "mild" severity).
* Subjects must have > or equal to 3 months of antipsychotic exposure.
* Other causes of involuntary movements have been ruled out.
* Psychiatrically stable as defined by outpatient status for > or equal to 2 months.
* No change in dopamine antagonist agent or dose for > or equal to 2 months or change in other prescribed medications for > or equal to 1 month prior to enrollment
* Patients must be 18-80 years of age.
* Patients must demonstrate adequate decisional capacity to make a choice about participating in this research study and must provide written informed consent to participate.
* Women who can become pregnant must be using an adequate method of contraception to avoid pregnancy throughout the study. Acceptable methods include oral, injectable or implanted contraceptives, intrauterine devices or barrier methods such as condoms, diaphragm and spermicides. Women who can become pregnant must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test at the Screening Visit.

Exclusion Criteria:

* Inpatient status
* Clinical Global Impression Severity (CGI-S) score > or equal to 6.
* Evidence of any medical condition(s) that could confound the presence of TD.
* Currently taking more than 2 antipsychotic medications.
* Currently taking levodopa.
* Current or prior treatment with valbenazine or deutetrabenazine within the past 3 months.
* Current or prior treatment with pyridoxine within the past 3 months.
* Women who are pregnant or breastfeeding.
* Alcohol use disorder as determined by the SCID within the past month.
* Substance use disorder (except caffeine and nicotine) as determined by the SCID within the past month.
* No serious and unstable medical condition(s) in the judgment of the investigator.
* DSM-V diagnosis of intellectual disability, moderate or greater severity; or diagnosis of major neurocognitive disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Mean Difference in AIMS scores | Baseline, Week 8
  Mean difference in Abnormal Involuntary Movement Scale (AIMS) total scores in participants assigned to pyridoxine and participants assigned to placebo from baseline to Week 8.
  The severity of TD symptoms is assessed by the Abnormal Involuntary Movement Scale (AIMS) total score (sum of items 1 through 7). The AIMS total dyskinesia score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.

SECONDARY OUTCOMES:
Mean Difference in Barnes Akathisia Rating Scale Scores | Baseline, Week 8
  Mean difference in Barnes Akathisia Rating Scale (BARS) scores in participants assigned to pyridoxine and participants assigned to placebo from baseline to Week 8.
  Barnes Akathisia Scale (BARS) is a rating scale that is administered by physicians to assess the severity of drug-induced akathisia, which is a movement disorder characterized by a feeling of inner restlessness and a compelling need to be in constant motion. The following subcategories are scored: objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness and are rated on a 4-point scale from 0 - 3. In addition, the global clinical assessment of akathisia uses a 6-point scale ranging from 0 - 5 (absent to severe). The total score ranges from 0 to 14 with a higher score indicating increased severity.
Mean Difference in Simpson Angus Scale Scores | Baseline, Week 8
  Mean difference in Simpson Angus Scale (SAS) scores in participants assigned to pyridoxine and participants assigned to placebo from baseline to Week 8.
  The Simpson-Angus Scale (SAS) is a 10-item testing instrument used to evaluate drug-related extrapyramidal syndromes. The following items are included in the SAS: gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella reflex, tremor, and salivation. Total score ranges from 0 to 40 with a higher score indicating increased severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lars F Jarskog, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Lerner V, Miodownik C, Kaptsan A, Cohen H, Matar M, Loewenthal U, Kotler M. Vitamin B(6) in the treatment of tardive dyskinesia: a double-blind, placebo-controlled, crossover study. Am J Psychiatry. 2001 Sep;158(9):1511-4. doi: 10.1176/appi.ajp.158.9.1511. PMID 11532741